CLINICAL TRIAL: NCT03962127
Title: MIDNOR-STROKE A Prospective Observation Study of a Cohort of 800 Patients With First Ever Ischemic Stroke in Central Norway
Brief Title: MIDNOR-STROKE- a Long Term Follow-up Study of Patients With First Ever Ischemic Stroke in Central Norway
Status: Active, not recruiting | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Helse Midt-Norge (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/453
Record Dates: First submitted 2019-05-17; First posted 2019-05-23 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Cardiovascular Diseases; Cardiovascular Risk Factor; Brain Ischemia; Cerebrovascular Disorders; Nervous System Diseases; Central Nervous System Lymphoma; Pathologic Processes; Vascular Diseases
Keywords: Cardiovascular risk factors; Risk Assessment; Severity of Illness Index; Mortality; Recurrent stroke; Health-related quality of life; modified Rankin scale; NIHSS; Fatigue severity score; Hospital anxiety and depression scale; Montreal cognitive assessment
MeSH Terms: conditions — Stroke; Cardiovascular Diseases; Brain Ischemia; Cerebrovascular Disorders; Nervous System Diseases; Pathologic Processes; Vascular Diseases; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First time ischemic stroke: Patients with a first event of ischemic stroke admitted to hospitals in Central Norway.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Annually 13000 Norwegians experience an ischemic stroke. The number of stroke is anticipated to increase with 50% within 2030 due to a growing number of elderly. Many of them will have severe function deficits and reduced quality of life. The investigators have established a cohort consisting of 800 patients with first time ischemic stroke treated at hospitals in Central Norway. The investigators want to study the incidence and prognostic markers for death, recurrent stroke and severe functional deficits during a period of 10 years after the initial ischemic stroke. The investigators want to focus on the impact of physical functioning, the level of physical activity and use of medication for secondary prevention on the incidence of death, recurrent stroke and severe functional deficits. The investigators are especially interested in the importance of fulfilling the treatment targets for blood pressure and cholesterol and the importance of smoking cessation in stroke survivors. Our objective is to improve todays stroke treatment and achieve a more efficient use of the health resources in order to increase survival after stroke maintaining a good physical and psychological function and quality of life.

DETAILED DESCRIPTION:
MIDNOR STROKE is a descriptive prospective longitudinal cohort study, which includes patients with a first event of ischemic stroke admitted to hospitals in Central Norway. The overall objective of this study is to complete a 10-year follow-up of patients with ischemic stroke.

Patient recruitment started 01.09.2015 and ended 01.11.2017. During this time-period, a total of 802 patients were recruited. Patient follow-up at 3 months is completed and follow-up at 12 months will be completed 01.11.18.

All participants met the following inclusion criteria; cerebral infarction according to ICD-10 CM code I63, > 18 years of age, first time stroke, resident in Central-Norway and recruited within a timeframe of 7 days of hospital admission. Patients were excluded if focal neurological symptoms turned out to be not stroke-related or if there were significant physical disabilities prior to stroke (defined as Modified Rankin ≥5)

Eligible stroke patients were recruited during acute stay in hospital. Written informed consent was obtained from all potential stroke patients and from their legal caretakers (mostly a close family member), admitted to the hospital and each subject signed an informed consent form. All participants were examined and treated in line with The Recommended Guidelines for treatment and rehabilitation of stroke, which includes clinical examinations, blood tests, assessment of risk profile and additional relevant examinations.

Stroke patients were recruited and patient data collected by a designated nurse during the initial stay at the hospital. Either a nurse or research assistant in the project performed patient follow-up at 3 and 12 months. Data collected at 3 months included data from a clinical and physical assessment, interview, questionnaires and medical records. Follow-up data at 12 months is collected by phone interview and questionnaires.

The data have been collected at baseline, 3 - and 12 months. Further data collection is planned at 3, 5 and 10 years.

The comprehensive data collection in MIDNOR STROKE at baseline includes data on pre-stroke function (Barthel index, Nottingham ADL, Modified rankin scale), life style risk factors, stroke severity (NIHSS, SSS, TOAST classifications), previous disease, vital signs (i.e. blood pressure, pulse, oxygen saturation), blood values, complications during hospital stay, medication and medical images during hospital stay. Assessment at 3 months included information on physical function, physical activity (HUNT - International physical activity questionnaire), cognitive function (Montreal cognitive assessment), depression (Hospital and anxiety and depression scale), fatigue (Fatigue severity score) and health related quality of life (EQ- 5D- 5L). Data collection at 12 months includes data on physical function, medication, depression, fatigue and health related quality of life.

Additional data will be collected from the Norwegian Stroke Registry, The Norwegian Patient registry, The Norwegian cardiovascular disease registry and The Norwegian Cause of Death registry.

The overall aim for MIDNOR STROKE is to establish a cohort of patients with first- time stroke to study the occurrence and predictors for recurrent stroke, mortality, physical activity, disability and the quality of life during a 10-year period.

MIDNOR STROKE contains six work packages, which address the key areas of interest in the project:

1. Recurrent stroke, mortality, disability and quality of life after stroke
2. Secondary prevention of stroke in relation to recurrent stroke, mortality, disability and quality of life.
3. Physical activity and function among stroke patients
4. Prediction models for recurrent stroke, disability and quality of life after stroke
5. Pathophysiologic mechanisms of acute ischemic stroke
6. Stroke health economics, health care resources cost and use

ELIGIBILITY:
Inclusion criteria:

* Cerebral infarction according to ICD-10 CM code I63
* > 18 years of age
* First time stroke resident in Central-Norway
* Recruited within a time frame of 7 days of hospital admission.

Exclusion criteria:

* Focal neurological symptoms turned out to be not stroke-related
* Significant physical disabilities prior to stroke (defined as Modified Rankin ≥5).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in a hospital in Central Norway for first time ischemic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of recurrent stroke after first ever ischemic stroke | 3 months
  Measured by using data from the Norwegian Stroke Registry and other Norwegian Cardiovascular registries including patient questionnaires
The incidence of recurrent stroke after first ever ischemic stroke | 1 year
  Measured by using data from the Norwegian Stroke Registry and other Norwegian Cardiovascular registries including patient questionnaires
The incidence of recurrent stroke after first ever ischemic stroke | 3 years
  Measured by using data from the Norwegian Stroke Registry and other Norwegian Cardiovascular registries including patient questionnaires
The incidence of recurrent stroke after first ever ischemic stroke | 5 years
  Measured by using data from the Norwegian Stroke Registry and other Norwegian Cardiovascular registries including patient questionnaires
The incidence of recurrent stroke after first ever ischemic stroke | 10 years
  Measured by using data from the Norwegian Stroke Registry and other Norwegian Cardiovascular registries including patient questionnaires
Mortality after first ischemic stroke | 3 months
  Measured with data from Norwegian Death Registry
Mortality after first ischemic stroke | 1 year
  Measured with data from Norwegian Death Registry
Mortality after first ischemic stroke | 3 years
  Measured with data from Norwegian Death Registry
Mortality after first ischemic stroke | 5 years
  Measured with data from Norwegian Death Registry
Mortality after first ischemic stroke | 10 years
  Measured with data from Norwegian Death Registry
Functional disability after stroke | 3 months after stroke
  Modified rankin scale 3 - 5 (the degree of disability, total range 0 - 6, value above 2 represents a worse outcome)
Functional disability after stroke | 1 year after stroke
  Modified rankin scale 3 - 5 (the degree of disability, total range 0 - 6,value above 2 represents a worse outcome)
Functional disability after stroke | 3 years after stroke
  Modified rankin scale 3 - 5 (the degree of disability, total range 0 - 6, value above 2 represents a worse outcome)
Functional disability after stroke | 5 years after stroke
  Modified rankin scale 3 - 5 (the degree of disability, total range 0 - 6, value above 2 represents a worse outcome)
Functional disability after stroke | 10 years after stroke
  Modified rankin scale 3 - 5 (the degree of disability, total range 0 - 6, value above 2 represents a worse outcome)
Health-related quality of life after stroke | 3 months after stroke
  EQ-5D-5L (5 Levels from 1-5 in 5 categories where values above 2 represents reduced life quality)
Health-related quality of life after stroke | 1 year after stroke
  EQ-5D-5L(5 Levels from 1-5 in 5 categories where values above 1 represents reduced life quality)
Health-related quality of life after stroke | 3 years after stroke
  EQ-5D-5L(5 Levels from 1-5 in 5 categories where values above 1 represents reduced life quality)
Health-related quality of life after stroke | 5 years after stroke
  EQ-5D-5L (5 Levels from 1-5 in 5 categories where values above 1 represents reduced life quality)
Health-related quality of life after stroke | 10 years after stroke
  EQ-5D-5L (5 Levels from 1-5 in 5 categories where values above 1 represents reduced life quality)

SECONDARY OUTCOMES:
Cost-benefit analysis | 1, 5 and 10 years
  Economic analysis that compares the costs of admission to hospital versus outpatient assessment of patients who have had transient ischemic attacks
Proportion of patients reaching secondary prevention targets | 3 months, 1, 3, 5 and 10 years
  Blood samples and questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bent Indredavik, PhD Prof, Study Director — Norwegian University of Science and Technology
Locations (8):
- Norway (8):
  - Ålesund Sykehus, Ålesund
  - Kristiansund Sykehus, Kristiansund
  - Levanger Sykehus, Levanger
  - Molde Sykehus, Molde
  - Namsos Sykehus, Namsos
  - Orkdal Sykehus, Orkanger
  - St Olavs Hospital, Trondheim
  - Volda Sykehus, Volda

IPD SHARING:
Plan to Share IPD: No